CLINICAL TRIAL: NCT07230678
Title: The Effect of an Environmentally Based Education Program on Adolescents' Environmentally Friendly Behaviors and Ecological Footprint Awareness: A Quasi-Experimental Study
Brief Title: The Effect of an Environmentally Based Education Program on Environmentally Friendly Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Busra Altinel, PhD, Selcuk University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 24202023
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Environmental Contamination; Environment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Environment-Based Education Program, consisting of three weeks and three sessions, was implemented for the intervention group students.
  Interventions: Behavioral: Environmentally Based Education Program
- Control (No Intervention): No intervention was implemented

INTERVENTIONS:
Behavioral: Environmentally Based Education Program — Week One: "Environment and Environmental Problems": The first week of the Environmentally Based Education Program aimed to equip participants with the skills to assess the causes of environmental problems and their potential consequences, as well as to help them develop solutions to combat environmental problems.
  Week Two: "Developing Environmentally Friendly Behaviors": The second week of the Environmentally Based Education Program aimed to assess what environmentally friendly behaviors are and what can be done to improve them.
  Week Three: "Ecological Footprint Awareness": The third week of the Environmentally Based Education Program aimed to evaluate the literal meaning of "ecological footprint" and what can be done to raise awareness on this issue.
  Arms: Intervention

SUMMARY:
This study was conducted to determine the effects of an environmentally-based education program implemented for adolescents on their environmentally friendly behaviors and ecological footprint awareness.

Research Hypotheses

Adolescents who received an environmentally-based education program aimed at developing environmentally friendly behaviors and increasing their ecological footprint awareness compared to the control group:

H1-0: There is no difference in terms of environmentally friendly behavior levels.

H2-0: There is no difference in terms of ecological footprint awareness levels. The Environment-Based Education Program, consisting of three weeks and three sessions, was implemented for the intervention group students.

ELIGIBILITY:
Inclusion Criteria:

* 10th grade students, ability to speak and understand Turkish

Exclusion Criteria:

* Previous environmental education, any communication skills, or a medically diagnosed mental illness

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Environmentally Friendly Behavior Scale | Week after intervention
  The scale, developed to determine participants' environmentally friendly behaviors, consists of a total of 26 items on a 5-point Likert-type scale ranging from 1 (Not at all) to 5 (A lot). The environmentally friendly behavior scale is rated as "26-46 points is very low," "47-67 points is low," "68-88 points is moderate," "89-109 points is high," and "110-130 points is very high."

SECONDARY OUTCOMES:
Ecological Footprint Awareness Scale | Week after intervention
  It aims to determine ecological footprint awareness levels. The scale consists of 46 questions across five subscales: food, transportation and shelter, energy, waste, and water consumption. The third item on the 5-point Likert-type scale is reverse-scored. As the score on the scale increases, so does the level of ecological footprint awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol